CLINICAL TRIAL: NCT01303757
Title: A Novel Diet-Phenotype Interaction Affecting Body Weight
Acronym: FRESH Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Broad Institute of MIT and Harvard (Other)
Responsible Party: Principal Investigator, David S. Ludwig, MD, PhD, Director, Obesity Prevention Center, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-04-0156
Record Dates: First submitted 2011-02-22; First posted 2011-02-25 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: obesity
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low glycemic load diet (Experimental): Low glycemic load diet
  Interventions: Behavioral: Dietary counselling
- Low fat diet (Active Comparator): Low fat diet
  Interventions: Behavioral: Dietary counselling

INTERVENTIONS:
Behavioral: Dietary counselling

SUMMARY:
The primary aim of the study is to examine insulin secretion as an effect modifier of the efficacy of a low-fat vs. low-glycemic load diet for weight loss among overweight/obese young adults in an 18-month, prospectively stratified, multi-center randomized controlled trial.

DETAILED DESCRIPTION:
In recent years, diets of widely varying composition have been used in the treatment of obesity. While none of these diets has produced consistent, long-term weight loss, some individuals on virtually all types of diets do remarkably well. One explanation for this variation among individuals is differences in motivation and behavior. However, underlying biological differences may also play an important role. Previous work has identified insulin secretion (as quantified by serum insulin concentration at 30 minutes following a standard 75-gram oral glucose load) as an important biological determinant. This randomized-controlled, multi-center trial aims to test the hypothesis that insulin secretion will predict which type of diet will work best for each individual. A total of 160 obese young adults (18 to 40 years) will be assigned to one of two diets: low-fat (60% carbohydrate, 20% fat, 20% protein) or low-glycemic load (45% carbohydrate, 35% fat, 20% protein). Participants will be enrolled at two sites (Children's Hospital Boston or University of North Carolina-Chapel Hill) and assigned to diet groups according to baseline insulin secretion status. The protocol will include an intensive 6-month intervention period and a 12-month follow-up period. Registered dietitians will provide nutrition education and behavioral counseling during group workshops and scheduled telephone calls. In an effort to avoid confounding, close attention will be paid to control for treatment intensity, physical activity prescriptions, and behavioral methods between groups. The primary endpoint will be percent body fat by DXA scan. Secondary endpoints will include cardiovascular and diabetes risk factors. Repeated, 24-hour dietary and physical activity recall interviews will provide process data. Metabolomic profiling and molecular analysis of identified metabolites will be conducted to characterize phenotype and explore potential physiological mechanisms. A successful outcome of this work will inform the practice of "personalized" nutritional therapy, enhancing the ability to select the most efficacious weight loss diet for an individual based on underlying biological differences.

ELIGIBILITY:
Inclusion Criteria

* Aged 18 to 40 years.
* Body mass index (BMI) ≥ 27 kg/m2.
* Body weight ≤ 300 lb.
* Access to a working telephone.
* Clearance in writing from a primary care provider (i.e., physician or nurse practitioner) to rule out pre-existing medical conditions.
* Willing and able to attend group workshops (for dietary intervention) on specified evenings.

Exclusion Criteria

* Physician diagnosis of a major medical illness or eating disorder.
* Chronic use of any medication that may affect study outcomes (e.g., insulin-sensitizing agents).
* Current smoking (i.e., 1 cigarette in the past week).
* Physical, mental, or cognitive handicaps that prevent participation.
* Another member of the family (i.e., first degree relative) or household participating in the study.
* Planning to relocate from current area of residence during the proposed timeframe for study participation.
* If female, planning to become pregnant during the 18 months of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percent body fat by dual-energy x-ray absorptiometry (DXA) | 18 months

SECONDARY OUTCOMES:
Triglyceride | 18 months
HDL cholesterol | 18 months
LDL cholesterol | 18 months
C-reactive protein | 18 months
Plasminogen Activator Inhibitor-1 | 18 months
Fasting blood glucose | 18 months
Insulin resistance | 18 months
Blood pressure | 18 months
Trunk fat | 18 months

OTHER OUTCOMES:
Serum insulin concentration 30 minutes following a standard 75-gram oral glucose load | 18 months
  Effect modification
Metabolomic profile | 18 months
  Effect modification
Insulin sensitivity | 18 months
  Effect modification
Abdominal-to-total fat ratio | 18 months
  Effect modification
Waist-to-hip ratio | 18 months
  Effect modification

CONTACTS AND LOCATIONS:
Overall Officials: Cara B Ebbeling, PhD, Study Director — Boston Children's Hospital; David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Leslie Fischer, PhD, Study Director — UNC Chapel Hill
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina